CLINICAL TRIAL: NCT03505541
Title: Effect of Adiponectin and TNFa on Uterine Contractility in GDM and Obese Pregnant Patients
Brief Title: Adipokines Effect in Myometrial Contractility
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00002972
Record Dates: First submitted 2018-04-12; First posted 2018-04-23 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Myometrium; Contractility; GDM; Obesity
MeSH Terms: conditions — Obesity | interventions — Adiponectin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Healthy, term, non-obese (BMI < 30) pregnant women with a singleton gestation scheduled for CS delivery at 37-41 weeks of gestation.
  Interventions: Biological: Adiponectin and TNFa
- Study group 1: Term pregnant, non-obese (BMI <30), diagnosed with gestational diabetes, scheduled for CS delivery between 37-41 weeks of gestation.
  Interventions: Biological: Adiponectin and TNFa
- Study group 2: Term pregnant, obese (BMI >30), non-diabetic and scheduled for CS delivery between 37-41 weeks of gestation
  Interventions: Biological: Adiponectin and TNFa

INTERVENTIONS:
Biological: Adiponectin and TNFa — Adiponectin and TNFa are adipokines. Will be added to the myometrial biopsies to investigate their effect on the force of contractility

SUMMARY:
Investigate the effect of two adipokines which are adiponectin and TNFa on the force of myometrial contractility in diabetic, non-obese pregnant women and obese, non-diabetic term pregnant women at the time of scheduled cesarean delivery

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients scheduled for a CS at 37-41 weeks of gestation at M Health Birth Place
* Participants age ≥18.
* Full informed consent able to be provided by the participant.

Exclusion Criteria:

* Patients undergoing general anesthesia for their CS.
* Pre-gestational DM, and DM diagnosed <24 weeks gestation.
* Patients unable to consent for themselves
* Multiple gestation

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant subjects undergoing a scheduled C-section delivery.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Effect on force of contractility | 24 hours
  Determine the effect of adiponectin and TNFa on the force of myometrial contractility in diabetic, non-obese pregnant women and obese, non-diabetic term pregnant women at the time of scheduled cesarean delivery

SECONDARY OUTCOMES:
Force of contractility between study groups | 24 hours
  Compare the force of myometrial contractility in study groups compared to control group (non-DM, non-obese term pregnant patients)
Progesterone effect in control group | 24 hours
  Investigate the anti-inflammatory properties of Progesterone (P4) and 17a-Hydroxyprogesterone (HPC) on Adiponectin induced myometrial contractility in control group

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Jacobs, MD, Principal Investigator — University of Minnesota
Locations (1):
- Fairview Hospital, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT03505541/Prot_000.pdf
  • Informed Consent Form (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT03505541/ICF_001.pdf